CLINICAL TRIAL: NCT04967326
Title: Role of Clinical Pharmacists in Epilepsy Management at a General Hospital in Vietnam: A Before-and-after Study
Brief Title: Role of Clinical Pharmacists in Epilepsy Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Principal Investigator, Pham Hong Tham, Clinical pharmacist, Gia Dinh People Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-2015/CN-HĐĐĐ
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy
Keywords: epilepsy; role of pharmacist; adverse drug reaction; antiepileptic drug; Vietnam
MeSH Terms: conditions — Epilepsy; Drug-Related Side Effects and Adverse Reactions | interventions — Anticonvulsants; Carbamazepine; Phenytoin; Valproic Acid

ARMS (1):
- Patients with epilepsy (Experimental): The therapies of patients with epilepsy were optimized using pharmacists' interventions, including medication consultation, dosage adjustment, medication switching/discontinuation, or combination therapy.
  Interventions: Drug: Optimizing therapy with antiepileptic drugs (carbamazepine, phenytoin, valproic acid)

INTERVENTIONS:
Drug: Optimizing therapy with antiepileptic drugs (carbamazepine, phenytoin, valproic acid)

SUMMARY:
Clinical pharmacists have an important role in inter-professional healthcare collaboration for epilepsy management. However, the pharmacy practices of managing epilepsy are still limited in Vietnam, deterring pharmacists from routine adjustments of antiepileptic drugs, which could decrease the patients' quality of life. This study aimed to assess the effectiveness of pharmacist interventions in epilepsy treatment at a Vietnamese general hospital.

DETAILED DESCRIPTION:
Phenytoin, carbamazepine, and valproic acid, which are among the first-generation AEDs, are prescribed in many countries around the world, including Vietnam. These agents have complicated pharmacokinetics, which may result in alterations in absorption, distribution, and metabolism. This means that, given the same dose, the serum concentration of each drug may vary between patients. The management of epilepsy, as a result, requires inter-professional collaboration to ensure therapeutic optimization. As healthcare professionals, clinical pharmacists play an important role in epilepsy management, which includes establishing a therapeutic drug monitoring (TDM) protocol, adjusting doses, monitoring ADRs, etc.

However, the clinical pharmacy practices in epilepsy management are quite limited in Vietnam. The treatment gap-the proportion of people with epilepsy who are not adequately treated-still remains very high, especially in rural areas (84.7%), which probably results from discontinuing the treatment or refusing to take medications. This shows a need for pharmacist consultations for patients with epilepsy and their family members, as they may be lack information about AEDs or motivation in controlling potential seizures. In addition, the adjustments of antiepileptic drugs by pharmacists are not routine procedures, nor are monitored for effectiveness in many Vietnamese hospitals. This lack of engagement threatens the patients' safety and decreases their quality of life. To address this issue, certain interventions are needed to enable pharmacists to manage patients with epilepsy more systematically. This study was therefore conducted to evaluate the effectiveness of pharmacist interventions in epilepsy treatment at a general hospital in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* were prescribed a monotherapy or polytherapy of phenytoin, carbamazepine, or valproic acid.
* were treated for more than one month.

Exclusion Criteria:

* were pregnant or breastfeeding women.
* had a history of alcoholism.
* had liver or renal disease.
* were using drugs known to have an influence on cytochrome P450 enzymes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with two seizures or less | One year from the start of the study
  Patients with two seizures or less in a year were categorized as having good control, whereas those who had more were considered to have poor control.

SECONDARY OUTCOMES:
Number of patients who maintained an optimized concentration of antiepileptic drugs | One year from the start of the study
  The targeted therapeutic ranges for carbamazepine, phenytoin, and valproic acid were 4-12 mg/L, 10-20 mg/L, and 50-100 mg/L, respectively.

REFERENCES:
- [Derived] Pham HT, Tran MH, Nguyen NQ, Tan Vo V, Tran MH. Role of clinical pharmacists in epilepsy management at a general hospital in Vietnam: a before-and-after study. J Pharm Policy Pract. 2021 Dec 20;14(1):109. doi: 10.1186/s40545-021-00394-9. PMID 34930487